CLINICAL TRIAL: NCT06386432
Title: Culturally-Tailored, Avatar-Led MHealth Intervention to Aid Smoking Cessation Among Sexual and Gender Minority Young Adults in New Mexico
Brief Title: EQQUAL-NM for the Promotion of Smoking Cessation in Sexual and Gender Minority Young Adults in New Mexico
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never opened to accrual and will not proceed due to lack of funding.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Cancer Institute Center to Reduce Cancer Health Disparities (Unknown); New Mexico State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RG1124189; NCI-2024-02453 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020404 (Other: Fred Hutch/University of Washington Cancer Consortium); U54CA132381 (NIH)
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-04

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Smoking Devices; Health Promotion; Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Any outcome evaluator who has contact with participants will remain blinded to treatment group assignment until the final set of questions regarding acceptability of specific program components is asked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (EQQUAL-NM, Program A) (Experimental): Participants receive self-guided smartphone app-delivered EQQUAL-NM (Program A) intervention on study. Participants also receive motivational messages, reminders and smoking cessation information via text messages. Some participants also complete at-home saliva sample collection during follow-up.
  Interventions: Behavioral: Smartphone App-delivered Smoking Cessation Intervention; Other: Health Promotion and Education; Other: Biospecimen Collection; Other: Questionnaire Administration
- Arm II (EQQUAL-NM, Program B) (Active Comparator): Participants receive self-guided smartphone app-delivered EQQUAL-NM (Program B) intervention on study. Participants also receive motivational messages, reminders and smoking cessation information via text messages. Some participants also complete at-home saliva sample collection during follow-up.
  Interventions: Behavioral: Smartphone App-delivered Smoking Cessation Intervention; Other: Health Promotion and Education; Other: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Smartphone App-delivered Smoking Cessation Intervention — Receive access to EQQUAL-NM (Program A) intervention
  Other Names: Smoking and Tobacco Use Cessation Intervention
  Arms: Arm I (EQQUAL-NM, Program A)
Behavioral: Smartphone App-delivered Smoking Cessation Intervention — Receive access to EQQUAL-NM (Program B) intervention
  Other Names: Smoking and Tobacco Use Cessation Intervention
  Arms: Arm II (EQQUAL-NM, Program B)
Other: Health Promotion and Education — Receive text message reminders, motivational messages and prompts via SMS text messages (Program A)
  Other Names: Text Message-Based Intervention
  Arms: Arm I (EQQUAL-NM, Program A)
Other: Health Promotion and Education — Receive text message reminders, motivational messages and prompts via SMS text messages (Program B)
  Other Names: Text Message-Based Intervention
  Arms: Arm II (EQQUAL-NM, Program B)
Other: Biospecimen Collection — Complete at-home saliva sample collection
  Other Names: Saliva Sample Collection
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial assesses the acceptability and efficacy of Empowered, Queer, Quitting, and Living--New Mexico (EQQUAL-NM), a smoking cessation intervention for sexual and gender minority young adults in New Mexico. Smoking prevalence among sexual and gender minority (SGM) adults in New Mexico is more than twice as high as non-SGM adults. Helping young adult tobacco users to quit is critical, yet there have been few efforts to develop tailored treatments specifically for this population. EQQUAL-NM is a digital smoking cessation intervention designed specifically for SGM young adult smokers in New Mexico and may help them quit smoking.

DETAILED DESCRIPTION:
OUTLINE:

Participants are randomized to 1 of 2 groups.

GROUP I: Participants receive access to a self-guided, smartphone app-delivered quit smoking program, called EQQUAL-NM (Program A) that helps explore personal values and teaches participants about smoking triggers and skills to help them manage cravings and accept thoughts and feelings related to smoking. Participants receive text message reminders and prompts on study. Some participants also undergo collection of a saliva sample during follow-up.

GROUP II: Participants receive access to a self-guided, smartphone app-delivered quit smoking program, called EQQUAL-NM (Program B) that is based on current clinical practice guidelines for tobacco cessation to help them quit smoking. This program helps with quit advice, tracking progress on quitting smoking, and managing cravings. Participants receive text message reminders and prompts on study. Some participants also undergo collection of a saliva sample during follow-up.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify being between 18 and 30 years of age
* Self-identify as a sexual and/or gender minority (i.e., a sexual orientation other than straight and/or gender that doesn't match sex assigned at birth)
* Currently reside in New Mexico, with a New Mexico mailing address, and anticipate remaining in New Mexico for the duration of the study (3 months)
* Self-report smoking at least 1 cigarette per week in the 30 days prior to screening
* Own an Android phone or iPhone
* Have at least weekly internet access for the next three months
* Willing and able to stream audio and video for this study
* Current use of a personal email account
* Current use of text messaging
* Interested in participating in the study for themselves (versus [vs] someone else)
* Self-report that they have not participated in one of Fred Hutch's/NMSU's prior smoking cessation studies
* Understand and agree to the conditions of compensation
* Currently not incarcerated
* Participants must be willing to use the assigned intervention program, complete the study assessments, and agree to the online consent form in English

Exclusion Criteria:

* Current use of other tobacco cessation treatments at the time of screening, including pharmacotherapy or behavioral support (but initiating these treatments during the study is allowed)
* Member of the same household as another research participant
* Previous use of the National Cancer Institute (NCI) QuitGuide app
* Google voice number as sole phone number
* Does not pass study fraud prevention protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Participant satisfaction | At 3-month follow-up
  Self-report of satisfaction overall and with specific program components will be rated on a 5-point Likert-type scale. Higher scale scores indicate higher satisfaction with the app.
Number of logins to the assigned application | Up to 3-month follow-up
  Server-recorded number of app openings over 3 months

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence (PPA) from all nicotine and tobacco products | At 3 months
  Self-report of no nicotine/tobacco product use over the previous 7 days, with the exception of FDA-approved medications
Biochemically confirmed 7-day point prevalence abstinence (PPA) from all nicotine/tobacco products | At 3 months
  Self-report of no nicotine/tobacco product use over the previous 7 days, with the exception of FDA-approved medications, biochemically confirmed via saliva cotinine
Self-reported 30-day PPA from all nicotine/tobacco products | At 3 months
  Self-report of no nicotine/tobacco product use over the previous 30 days, with the exception of FDA-approved medications
Biochemically confirmed 30-day PPA from all nicotine/tobacco products | At 3 months
  Self-report of no nicotine/tobacco product use over the previous 30 days, with the exception of FDA-approved medications, biochemically confirmed via saliva cotinine
Self-reported 7-day PPA from cigarette smoking | At 3 months
  Self-report of no cigarette smoking over the previous 7 days
Self-reported 30-day PPA from cigarette smoking | At 3 months
  Self-report of no cigarette smoking over the previous 30 days
Change in Contemplation Ladder scores | At baseline and at 3-month follow-up
  Contemplation Ladder scores will be used to assess readiness to quit using cigarettes. Ladder scores are on a 0 to 10 scale, with higher change scores meaning greater increases readiness to quit.
Change in acceptance of tobacco-use triggers | At baseline and at 3-month follow-up
  Change in acceptance of tobacco-use triggers will be measured using the Avoidance and Inflexibility Scale. Higher change scores indicate greater improvement in acceptance of tobacco use triggers.
Change in values-guided action | At baseline and at 3-month follow-up
  Change in values-guided action measured using the Values Questionnaire. Higher change scores indicate greater improvement in values-guided action.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimee Heffner, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No